CLINICAL TRIAL: NCT04619030
Title: Augmented Reality (AR): The Future of "Patient Information Leaflets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: The Glasgow School of Art (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: GN19HS442
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Sarcoma; Breast Cancer; Cleft Lip and Palate; Surgical Flap
Keywords: patient information leaflet; augmented reality
MeSH Terms: conditions — Sarcoma; Breast Neoplasms; Cleft Lip

STUDY DESIGN:
Intervention Model Description: Randomised crossover
Who Masked: Investigator, Outcomes Assessor
Masking Description: It is not possible to blind participants to visual information in the patient leaflet (augmented reality versus traditional). The data collected will be fully anonymised before statistical assessment by an independent statistical service
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Reality Leaflet (Experimental): Patient Leaflet with Augmented reality component
  Interventions: Other: Augmented Reality
- Traditional Leaflet (Active Comparator): Traditional leaflet without Augmented Reality component
  Interventions: Other: Traditional leaflet

INTERVENTIONS:
Other: Augmented Reality — The patient leaflet has an Augmented Reality model that appears out of the leaflet when viewed with a smartphone
  Arms: Augmented Reality Leaflet
Other: Traditional leaflet — Traditional leaflet with no Augmented Reality capability
  Arms: Traditional Leaflet

SUMMARY:
This project aims to assess a new type of Augmented Reality Patient Information leaflet, in order to demonstrate that it is a beneficial information resource to patients when facing the diagnosis of sarcoma, breast cancer or to explain difficult concepts such as cleft lip repair. There are no published studies on the use of AR in patient leaflets.

DETAILED DESCRIPTION:
At present, the traditional approach to patient education regarding diseases such as a new cancer diagnosis, is the patient information leaflet. Patient information leaflets often fail to convey the required medical information due to poor levels of literacy in the population, with 20% patients in the UK having the lowest level of adult literacy (equivalent to an individual who is unable to determine how much medicine to give a child from information printed on the package). "Health literacy" - the ability to obtain, understand, act on and communicate health information - is even lower, with estimates that 40% of patients have inadequate levels of health literacy. Additionally, there is a large knowledge gap between what doctors perceive patients understand about an illness, medication, or operation, and what patients actually comprehend and retain during consultation.

The plethora of problems of inadequate information, poor health literacy and patient-doctor knowledge disconnect, may be addressed with an approach to patient information leaflets using a platform that is entirely simulative and visual, thereby overcoming the problem of health literacy. The study builds upon pilot work by this research team on patient leaflets using AR to aid in patient education, visualisation and retention of information (Lo et al 2019).

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone reconstructive surgery
* patients who are awaiting reconstructive surgery
* patients with sarcoma
* patients with breast cancer
* patients with reconstructive flaps
* patients with or parents of patients with cleft lip and palate
* Patients with dyslexia will be included

Exclusion Criteria:

* Cannot speak or read English
* Blind/severely visually impaired

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Mental Effort Rating Scale | Single point at day 1 (Patient assesses leaflet once after reading leaflet)
  Validated scale for cognitive load/ ease of understanding leaflet. Single item scale with rating 1 = very, very low mental effort to 9 = very, very high mental effort. Lower score is better

SECONDARY OUTCOMES:
Overall Patient Satisfaction | Single point at day 1 (Patient assesses leaflet once after reading leaflet)
  Visual analogue scale, overall satisfaction with patient leaflet. Visual analogue scale will be converted to numerical scale 0-100, with higher being better or more satisfied
Instructional Motivation Materials Survey | Single point at day 1 (Patient assesses leaflet once after reading leaflet)
  Assessment of patient learning motivation after reading leaflet. 36 items, each item rated by Likert scale 1-5. Higher score is better.
Usefulness Scale for Patient Information (USE scale) | Single point at day 1 (Patient assesses leaflet once after reading leaflet)
  9 item scale with Likert rating 0-10 for each item. Total score out of 90, with 3 sub scales measuring cognitive, emotional and behavioural dimensions. Higher score is better.

OTHER OUTCOMES:
Subjective interview | Single point at day 1 (Patient assesses leaflet once after reading both leaflets)
  Patients will be interviewed regarding opinions of the two types of patient leaflet.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Canniesburn Regional Plastic Surgery and Burns Unit, Glasgow, Scotland
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Royal Hospital for Children, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Available on reasonable written request following publication.
Supporting Information: Study Protocol
Time Frame: Following publication and for 1 year
Access Criteria: Available on reasonable written request

REFERENCES:
- [Derived] Lo SJ, Chapman P, Young D, Drake D, Devlin M, Russell C. The Cleft Lip Education with Augmented Reality (CLEAR) VR Phase 2 Trial: A Pilot Randomized Crossover Trial of a Novel Patient Information Leaflet. Cleft Palate Craniofac J. 2023 Feb;60(2):179-188. doi: 10.1177/10556656211059709. Epub 2022 Jan 4. PMID 34982018